CLINICAL TRIAL: NCT01157572
Title: Effect of Beta Blockade on Left Ventricular Remodeling and Function in Moderate to Severe Asymptomatic Aortic Regurgitation
Acronym: BAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Ghent (Other); University Hospital, Gentofte, Copenhagen (Other); University Hospital, Akershus (Other); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Stig Urheim, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUDRACTNR: 2007-000518-34
Record Dates: First submitted 2010-07-05; First posted 2010-07-07 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Aortic Valve Insufficiency
Keywords: Aortic valve insufficiency; Beta-blocker
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoprolol (Active Comparator)
  Interventions: Drug: Metoprolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoprolol — Patients with moderate to severe aortic valve insufficiency will be randomized to Metoprolol
  Arms: Metoprolol
Drug: Placebo — Patients with moderate to severe aortic valve insufficiency will be randomized to Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of beta-blocker on left ventricular (LV) remodeling in asymptomatic patients with moderate to severe aortic regurgitation.

DETAILED DESCRIPTION:
The left ventricle responds to the volume load of chronic aortic regurgitation (AR) with a series of compensatory mechanisms, including an increase in end-diastolic volume, an increase in chamber compliance that accommodates the increased volume without an increase in filling pressures, and a combination of eccentric and concentric hypertrophy. The greater diastolic volume permits the ventricle to eject a large total stroke volume to maintain forward stroke volume in the normal range. This is accomplished through rearrangement of myocardial fibers with the addition of new sarcomeres and development of eccentric LV hypertrophy. As a consequence left ventricular ejection fraction will remain in the normal range.

The clinical course of chronic aortic regurgitation is characterized by a prolonged phase of stability during which the left ventricle adapts to the volume overload. Eventually myocardial failure ensues through a series of complex events that include changes in myocyte phenotype due to re-expression of fetal genes, cellular apoptosis alteration in the expression and function of contractile proteins and changes in the extracellular matrix.

The role of long-term vasodilator therapy in the care of asymptomatic patients with severe aortic regurgitation is controversial. Vasodilator therapy has been used to reduce the regurgitant volume, afterload, left ventricular volumes, and wall stress in an effort to preserve left ventricular function and reduce left ventricular mass. Thus time to surgical intervention has been found to be delayed by calcium antagonists, ACE-inhibitors and hydralazine, while a more recent study did not find any effect of nifedipine or enalapril on time to surgery or left ventricular volume and function.

The decision to recommend operative intervention to the asymptomatic patient with chronic, severe aortic regurgitation (AR) is very difficult because aortic valve replacement (AVR) continues to entail immediate risk, and biologic and mechanical valves still have problems resulting in significant morbidity and mortality. On the other hand, the mortality rate in asymptomatic patients with AR is very low, and surgery does not improve the quality of life. Thus, the indication in asymptomatic patients must be delayed until changes occur that will predict an increased risk of operative or long-term death after AVR. At present indication for aortic valve replacement is development of symptoms, an increase in left ventricular volume or a decline in left ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe aortic valve insufficiency
* Asymptomatic

Exclusion Criteria:

* Arrhythmia
* Other severe valve disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Left ventricular end-diastolic volume | 6 months

SECONDARY OUTCOMES:
Left ventricular end-systolic volume | 6 months

REFERENCES:
- [Derived] Broch K, Urheim S, Lonnebakken MT, Stueflotten W, Massey R, Fossa K, Hopp E, Aakhus S, Gullestad L. Controlled release metoprolol for aortic regurgitation: a randomised clinical trial. Heart. 2016 Feb;102(3):191-7. doi: 10.1136/heartjnl-2015-308416. Epub 2015 Dec 9. PMID 26661319